CLINICAL TRIAL: NCT03675945
Title: Smartphone Evaluation of Postoperative Pain Profiles Following General Surgery in Children : a French Multi Center Randomized Trial (AlgoDARPEF)
Brief Title: Smartphone Evaluation of Postoperative Pain Profiles Following General Surgery in Children
Acronym: AlgoDARPEF
Status: Completed | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 18-HPNCL-05
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-07

CONDITIONS: Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pain is common following surgery in children. Currently, no recent review of pain profiles at home has been performed on pediatric population in France following general surgery in children. The aim of this study is to evaluate the duration and severity of pain felt by children using a mobile phone application. All children operated in the different centers and leaving home will be included in the study. Children's pain scores will be measured using PPMP-SF scale (Postoperative Pain Measure for Parents Short Form). Data on prescribed and administered analgesia, nausea-vomiting, behavioral problems and parental satisfaction will be collected. The expected results are an inventory's objective observation of postoperative pain profiles at home following the different pediatric surgeries in France. The study will also highlight the different risk factors of postoperative pain (type of surgery, parental causes, reasons due to the child, medical causes).

DETAILED DESCRIPTION:
Data from literature suggest that control of postoperative pain remains difficult and insufficient despite interventions to improve the management of children's home-based postoperative pain. In 2017, a recent Australian prospective audit confirms that pain is still underestimated and under-treated by medical staff and home-based families. Currently, no recent review of pain profiles at home has been performed on the pediatric population in France following general surgery in children. The aim of this study is to evaluate the duration and severity of pain felt by children using a mobile phone application.

The study is an epidemiological, observational, prospective and multicenter trial. All children operated in the different centers and leaving home will be included in the study. The peri-operative analgesic treatment will be left to the discretion of the various centers. In addition to the surgical follow-up, post-operative follow-up at home will be carried out using the smartphone application for all patients.

The use of the application will have been explained during the intervention's programming. The application will be downloaded by the parents at home. Parents will be alerted by notifications when they have tracking data to enter. The primary endpoint will be the evaluation of postoperative pain thanks to PPMP-SF scale. Data on prescribed and administered analgesia, nausea-vomiting, behavioral problems and parental satisfaction will be collected.

Statistical analysis will first include a descriptive study of the population. Qualitative data will be expressed as means and standard deviations, and quantitative data as numbers and percentages. Before carrying out each comparative analysis, the application's conditions of the tests used will be verified. The different tests will be considered significant at the 5% threshold unless otherwise specified.

The expected results are an inventory's objective observation of postoperative pain profiles at home following the different pediatric surgeries in France. The study will also highlight the different risk factors of postoperative pain (type of surgery, parental causes, reasons due to the child, medical causes).

A recent study in Sweden in adult population has shown that systematic e-assessment can improve patients' quality of recovery.

A mobile phone application on postoperative pain assessment in pediatric population would improve the management of children's pain and therefore improve the quality of postoperative recovery at home.

ELIGIBILITY:
Inclusion Criteria:

* All children operated in the centers participating in the study, regardless of age.
* Possession of a smartphone by one of the two parents.
* Affiliated parent or beneficiary of a Social Security scheme.
* Collection of the non-opposition of one of the parents or the representative of the parental authority

Exclusion Criteria:

* Parents who refused or do not understand the protocol
* Parents who don't have the necessary hardware to download the application for mobile phone
* Non-French parents
* Vulnerable people according to article L1121-6 of the public health code

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children operated in the different centers and leaving home will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 1576 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain's evaluation by parents | from day 0 until day 10
  Measure of pain with scale Postoperative Pain Measure for Parents Short Form (PPMP-SF) using the mobile phone application. PPMP-SF scale has 10 items about child behavior. Each item score is 0 or is 1, score of 0 equals an absent sign, score of 1 equals a present sign. Total score is 10. Significant pain is greater than or equal to 6.
Postoperative pain's evaluation by patients | from day 0 until day 10
  Measure of pain with auto-evaluation Visual Analog Scale (VAS), using mobile phone application. VAS score goes from 0 to 10. Significant pain is greater than or equal to 3.

SECONDARY OUTCOMES:
Evaluation of Pre-operative anxiety of parents | at the day before surgery
  Measure of parent Pre-operative anxiety by a visual analog scale using mobile phone application. Score goes from 0 to 10. Score of 0 equals no anxiety. Significant anxiety is greater than or equal to 3.
Evaluation of Pre-operative anxiety of 7 years old and over patients | at the day before surgery
  Self-evaluation of pre-operative anxiety with visual scale using mobile phone application. Score goes from 0 to 10. Score of 0 equals no anxiety. Significant anxiety is greater than or equal to 3.
measure of postoperative adverse events | from day 0 to day 10
  count of post-surgery events : vomiting, nausea, medical visit using a questionary of mobile phone application

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Walrave, MD, Principal Investigator — Fondation Lenval - Nice Children Hospital CHU-Lenval
Locations (1):
- Hôpitaaux Pédiatriques de Nice CHU-Lenval, Nice, France

REFERENCES:
- [Derived] Walrave Y, Carles M, Evain JN, Ikonomoff T, Marie A, Ludot H, Bourdaud N, Kern D, Lejus-Bourdeau C, Orliaguet G, Rosello O, Ecoffey C, Savoldelli C, Perissier C, Delacquis M, Vare B, Donzeau D, Cousin C, Langlais E, Breaud J, Jonckheer K, Dadure C, De la Briere F; Association of French Pediatric Anaesthesia and Intensive Care Medicine (ADARPEF). A follow-up of pain reported by children undergoing outpatient surgery using a smartphone application: AlgoDARPEF multicenter descriptive prospective study. Pain. 2022 Nov 1;163(11):2224-2231. doi: 10.1097/j.pain.0000000000002620. Epub 2022 Mar 1. PMID 35239543